CLINICAL TRIAL: NCT07321080
Title: The Experience of Nociceptive and Neuropathic Pain: Differences in Levels of Central Sensitization
Brief Title: Central Sensitisation in Nociceptive and Neuropathic Pain
Acronym: ALGOS
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Anna Anselmo, Psychologist, IRCCS Centro Neurolesi Bonino Pulejo
Other Study IDs: CEL/U138/25
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Nociceptive Pain; Neuropathic Pain; Mixed Pain (Nociceptive and Neuropathic)
Keywords: CHRONIC PAIN; CENTRAL SENSITIZATION; NEUROPATHIC PAIN; NOCICEPTIVE PAIN; MIXED PAIN; LASER-EVOKED POTENTIALS; NEUROPSYCHOLOGICAL ASSESSMENT
MeSH Terms: conditions — Chronic Pain; Nociceptive Pain; Neuralgia | interventions — Neuropsychological Tests; Laser-Evoked Potentials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nociceptive pain: Patients suffering from nociceptive pain
  Interventions: Behavioral: Neuropsychological assessment; Behavioral: Laser evoked potentials
- Mixed pain: Patients suffering from mixed pain
  Interventions: Behavioral: Neuropsychological assessment; Behavioral: Laser evoked potentials
- Neuropathic pain: Patients suffering from neuropathic pain
  Interventions: Behavioral: Neuropsychological assessment; Behavioral: Laser evoked potentials

INTERVENTIONS:
Behavioral: Neuropsychological assessment — Neuropsychological assessment Standardized and ad hoc test battery for comprehensive neuropsychological assessment
Behavioral: Laser evoked potentials — Laser evoked potentials

SUMMARY:
This study aims to investigate differences in central sensitization among patients with chronic nociceptive pain, neuropathic pain, and mixed pain conditions. Chronic pain is a complex and multidimensional phenomenon involving sensory, cognitive, emotional, and behavioral components, often sustained by mechanisms of central sensitization that contribute to pain persistence and treatment resistance.

Using a multidimensional assessment approach, the study integrates self-report questionnaires, neuropsychological evaluation, psychological measures, treatment adherence assessment, and neurophysiological investigation through laser-evoked potentials (LEP). Participants will be evaluated at baseline and after 12 months to explore differences between pain types and longitudinal changes in central sensitization, cognitive functioning, emotional status, and engagement with treatment.

The findings are expected to improve the understanding of neurobiological and psychosocial mechanisms underlying different chronic pain phenotypes and to support more personalized and effective pain management strategies.

DETAILED DESCRIPTION:
This is an observational, prospective, longitudinal cohort study designed to examine central sensitization and its multidimensional correlates in patients with chronic pain. The study will be conducted at the IRCCS Centro Neurolesi "Bonino-Pulejo", P.O. "Piemonte", Messina, Italy.

The study population consists of adult patients (18-90 years) suffering from chronic pain and referred to the pain outpatient clinic or hospitalized in pain therapy units. Based on standardized screening instruments for pain classification (Douleur Neuropathique en 4 Questions - DN4 and PainDETECT Questionnaire - PD-Q), participants will be stratified into three cohorts: nociceptive pain, neuropathic pain, and mixed pain. The mixed group includes patients with overlapping nociceptive and neuropathic features or pain conditions that are not clearly classifiable within a single category, including nociplastic pain mechanisms.

All participants will undergo a comprehensive evaluation at baseline (T0) and at 12-month follow-up (T1). The assessment protocol includes measures of pain intensity and central sensitization (Numeric Pain Rating Scale, Central Sensitization Inventory), neurophysiological assessment of nociceptive pathways using laser-evoked potentials (LEP), cognitive screening (Montreal Cognitive Assessment), psychological status (Beck Depression Inventory and State-Trait Anxiety Inventory), pain-related self-efficacy (Pain Self-Efficacy Questionnaire), treatment engagement (Patient Health Engagement Scale), and medication adherence (Morisky Medication Adherence Scale).

Participants will also be stratified according to their pharmacological treatment at baseline, including non-steroidal anti-inflammatory drugs, paracetamol, opioids, cannabinoids, anticonvulsants/gabapentinoids, antidepressants, topical agents, and combination therapies. Changes in treatment during the follow-up period will be documented.

The primary objective is to compare levels of central sensitization among nociceptive, neuropathic, and mixed pain groups using both subjective (CSI) and objective (LEP) measures. Secondary objectives include the characterization of cognitive, psychological, and behavioral profiles associated with each pain type and the evaluation of longitudinal changes over time.

This multidimensional and longitudinal approach aims to clarify the role of central sensitization across different chronic pain phenotypes and to support more tailored and integrated therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Presence of chronic pain
* Diagnosis of nociceptive pain, neuropathic pain, mixed pain, or nociplastic pain
* Patients referring to the pain outpatient clinic
* Patients hospitalized in pain therapy units
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Presence of severe psychiatric disorders
* Presence of severe neurological disorders
* Presence of oncological diseases in terminal stage

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size was estimated using G*Power 3.1 based on the primary outcome measure, the Central Sensitization Inventory (CSI). A one-way ANOVA (omnibus test) comparing three groups (nociceptive pain, neuropathic pain, and mixed pain) with equal allocation (1:1:1) was assumed. The calculation was performed using a moderate effect size (f = 0.25), a two-sided significance level of α = 0.05, and a statistical power of 0.80.
  Based on these parameters, a minimum sample size of 159 participants was required (53 participants per group). Considering an expected dropout rate of approximately 15% over the 12-month follow-up period, the target enrollment was increased to approximately 185 participants, corresponding to about 62 participants per group.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
neuropsychological assessment | 24 months
  neuropsychological assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Centro Neurolesi Bonino Pulejo, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No